CLINICAL TRIAL: NCT04207034
Title: Effect of the Diode Laser on Bacteremia Associated With Periodontal Flap Surgery: A Clinico-Microbiological Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, proffesor/ Head of the department Periodontology, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_91549
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: The study was performed according to split- mouth design, and all teeth in the mouth were treated randomly using either the left or the right side of the maxilla and mandible for control , and the opposite side for the therapy. Each patient was entered into a clinical protocol consisting of two different treatment modalities.
  Group I (n=10) - Test group ( diode laser + flap surgery) Group II (n=10) - control group (flap surgery)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (investigator and outcome Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flap surgery and diode laser (Experimental): Patient will be asked to rinse with 0.2% chlorhexidine mouthwash. Following the administration of local anaesthesia 2% lignocaine hydrochloride ( with 1: 80,000 epinephrine) , Laser application will be carried out , with the help of 810 nm (A.R.C LASER FoxTM) diode laser with a flexible optic tip of 300µm . The sulci will be lased with a repeated beam ( 0.2 sec on 0.3 sec off) at an output power of 1.0 W.
  Intracrevicular incision will be placed with the help of 15c Bard Parker surgical blade , full thickness mucoperiosteal flap will be elevated .
  Debridement of granulation tissue will be done and flap will be suture back in position using 3-0 black breaded silk suture, the site will be covered with non eugenol periodontal dressing for protection.
  Postoperative instructions will be given to the patient. 2 ml blood will be collected at baseline(sample 1) , at 5 minutes (sample 2) and within 20-30 minutes (sample 3) of starting the procedure.
  Interventions: Procedure: flap surgery with diode laser
- flap surgery (Active Comparator): Patient will be asked to rinse with 0.2% chlorhexidine mouthwash. Following the administration of local anaesthesia 2% lignocaine hydrochloride ( with 1:80,000 epinephrine) ,intracrevicular incision will be placed with the help of 15c Bard Parker surgical blade , full thickness mucoperiosteal flap will be elevated .
  Debridement of granulation tissue will be done and flap will be suture back in position using 3-0 black breaded silk suture, the site will be covered with non eugenol periodontal dressing for protection.
  Postoperative instructions will be given to the patient. 2 ml blood will be collected at baseline(sample 1) , at 5 minutes (sample 2) and within 20-30 minutes (sample 3) of starting the procedure
  Interventions: Procedure: flap surgery

INTERVENTIONS:
Procedure: flap surgery with diode laser — Patient will be asked to rinse with 0.2% chlorhexidine mouthwash. Following the administration of local anaesthesia 2% lignocaine hydrochloride ( with 1: 80,000 epinephrine) , Laser application will be carried out , with the help of 810 nm (A.R.C LASER FoxTM) diode laser with a flexible optic tip of 300µm . The sulci will be lased with a repeated beam ( 0.2 sec on 0.3 sec off) at an output power of 1.0 W.
  Intracrevicular incision will be placed with the help of 15c Bard Parker surgical blade , full thickness mucoperiosteal flap will be elevated .
  Debridement of granulation tissue will be done and flap will be suture back in position using 3-0 black breaded silk suture, the site will be covered with non eugenol periodontal dressing for protection.
  Postoperative instructions will be given to the patient. 2 ml blood will be collected at baseline(sample 1) , at 5 minutes (sample 2) and within 20-30 minutes (sample 3) of starting the procedure.
  Arms: flap surgery and diode laser
Procedure: flap surgery — Patient will be asked to rinse with 0.2% chlorhexidine mouthwash. Following the administration of local anaesthesia 2% lignocaine hydrochloride ( with 1:80,000 epinephrine) ,intracrevicular incision will be placed with the help of 15c Bard Parker surgical blade , full thickness mucoperiosteal flap will be elevated .
  Debridement of granulation tissue will be done and flap will be suture back in position using 3-0 black breaded silk suture, the site will be covered with non eugenol periodontal dressing for protection.
  Postoperative instructions will be given to the patient. 2 ml blood will be collected at baseline(sample 1) , at 5 minutes (sample 2) and within 20-30 minutes (sample 3) of starting the procedure
  Arms: flap surgery

SUMMARY:
The objective of the present study is

1. To study the incidence and magnitude of bacteremia after periodontal flap surgery .
2. To compare and evaluate the effect of diode laser on frequency of bacteremia associated with periodontal flap surgery .
3. To study the incidence of bacteremia after laser therapy

DETAILED DESCRIPTION:
SOURCE OF DATA Patient visiting the Outpatient Section of the Department of Periodontology, Krishnadevaraya College of Dental Sciences and Hospital will be screened and randomly recruited for the study as per inclusion and exclusion criteria. The eligible subjects will be informed of the nature and benefits of the participation of the study and a written signed consent will be obtained. The study population will consist of twenty (n=20) subjects who will be age (30 to 40 years) and sex matched.

Sample Size The study was performed according to split- mouth design, and all teeth in the mouth were treated randomly using either the left or the right side of the maxilla and mandible for control , and the opposite side for the therapy. Each patient was entered into a clinical protocol consisting of two different treatment modalities.

Group I (n=10) - Test group ( diode laser + flap surgery) Group II (n=10) - control group (flap surgery)

SURGICAL PROCEDURE GROUP I (TEST GROUP) Patient will be asked to rinse with 0.2% chlorhexidine mouthwash. Following the administration of local anaesthesia 2% lignocaine hydrochloride ( with 1: 80,000 epinephrine) , Laser application will be carried out , with the help of 810 nm (A.R.C LASER FoxTM) diode laser with a flexible optic tip of 300µm . The sulci will be lased with a repeated beam ( 0.2 sec on 0.3 sec off) at an output power of 1.0 W.

Intracrevicular incision will be placed with the help of 15c Bard Parker surgical blade , full thickness mucoperiosteal flap will be elevated .

Debridement of granulation tissue will be done and flap will be suture back in position using 3-0 black breaded silk suture, the site will be covered with non eugenol periodontal dressing for protection.

Postoperative instructions will be given to the patient. 2 ml blood will be collected at baseline(sample 1) , at 5 minutes (sample 2) and within 20-30 minutes (sample 3) of starting the procedure.

GROUP II (CONTROL GROUP) Patient will be asked to rinse with 0.2% chlorhexidine mouthwash. Following the administration of local anaesthesia 2% lignocaine hydrochloride ( with 1:80,000 epinephrine) ,intracrevicular incision will be placed with the help of 15c Bard Parker surgical blade , full thickness mucoperiosteal flap will be elevated .

Debridement of granulation tissue will be done and flap will be suture back in position using 3-0 black breaded silk suture, the site will be covered with non eugenol periodontal dressing for protection.

Postoperative instructions will be given to the patient. 2 ml blood will be collected at baseline(sample 1) , at 5 minutes (sample 2) and within 20-30 minutes (sample 3) of starting the procedure

Collection of blood samples Six millilitres (6 ml) of blood samples will be drawn from the patient through an antecubital vein using strict aseptic technique via a 22- gauge sterile plastic cannula and sent for for qPCR analysis to quantify total bacterial load.

PCR ANALYSIS The polymerase chain reaction (PCR) is a laboratory technique for DNA replication that allows the "target" DNA sequence to be selectively amplified. The PCR involves the primer mediated enzymatic amplification of DNA. In this study Quantitive polymerase chain reaction is done.

* DNA from the blood samples will be extracted using the QIAamp DNA Blood Mini Kit according to the manufacture's recommendations.
* In order to quantify the total bacterial load, qPCR will be carried out using a universal primer to the 16S ribosomal RNA gene.
* Analysis was performed in a total volume of 6 ml blood.
* Samples for qPCR will be dispensed into well plates, sealed and centrifuged.
* Amplification will be done , settings for qPCR will be as follows: 95 degree centigrade for 10 minutes followed by 40 amplification cycles at 95 degree centigrade for 1 minute, 52 degree centigrade for 1 minute , 72 degree centigrade for 1 minute.
* After each cycle , PCR products will be monitored for the increase in fluorescence of SYBR green.
* All measurements will be performed in triplicate for both test and controls.
* For the negative control , ultrapure water will be used replacing the clinical sample.
* To determine the specificity of the amplified products, a melting curve will be obtained from 60 degree centigrade to ninty five degree centigrade, with continuous florescence measurement at each 1% increase in temperature.
* Data acquisition and analysis will be performed using the ABI 7500 software.

Statistical analysis Data will be subjected for normality test. Best on the data parametric or non parametric test will be performed. P value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with age 30 -40 years .
2. Systemically healthy patients.
3. Patients having probing depth of ≥ 5mm and ≤ 8 mm at minimum of two sites and good level of oral hygiene after initial therapy.
4. No signs of gingival inflammation

Exclusion Criteria:

1. Patient with history of smoking, antibiotic therapy within the previous three months.
2. Patient with subgingival restorations and use of antiseptic mouthwash.
3. Congenital or acquired cardiac defects, cardiac prosthesis.
4. Hematological disorder.
5. Immunocompromised patients

   -

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of bacteremia using PCR | After 24 hours of collection
  Bacteremia in venous blood before starting the procedure, after 5 minutes and within 30 minutes of the start of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Akanksha Dubey, MDS, Principal Investigator — Rajiv Gandhi University of Health Sciences; MLV Prabhuji, MDS, Study Director — Rajiv Gandhi University of Health Sciences
Locations (1):
- MLV Prabhuji, Bangalore, Karnataka, India